CLINICAL TRIAL: NCT03025022
Title: An Open-Label Study to Investigate the Absorption, Distribution, Metabolism, and Excretion of 14C-JNJ-42847922 After a Single Oral Dose of 40 mg in Healthy Subjects
Brief Title: A Study to Investigate the Absorption, Distribution, Metabolism, and Excretion of 14C-JNJ-42847922 After a Single Oral Dose of 40 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108268; 42847922EDI1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- 14C-JNJ-42847922 40 miiligram (mg) (Experimental): Participants will receive a single 40 mg oral dose of 14C-JNJ-42847922 on Day 1.
  Interventions: Drug: 14C-JNJ-42847922 40 mg

INTERVENTIONS:
Drug: 14C-JNJ-42847922 40 mg — Participants will receive a single 40 mg oral dose of 14C-JNJ-42847922 containing maximally 100 MicroCurie as a 40 milliLitre (mL) solution.

SUMMARY:
The objective of this study is to evaluate the absorption, distribution, metabolism, and excretion (ADME) of 14C-JNJ-42847922 in healthy subjects after a single oral dose of 40 milligram (mg) 14C-JNJ-42847922 containing maximally 100 MicroCurie. Safety and tolerability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they (healthy participants) understand the purpose of and procedures required for the study and are willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in the protocol
* Women may be eligible to participate if they are of non child-bearing potential, which is defined as (a) Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level (more than [>] 40 International Units Per Litre [IU/L] or milli-International Units per milliliter [mIU/mL]) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient; OR (b) Permanently Sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy
* Body mass index (BMI; weight kilogram [kg]/height^2 (meter [m]^2)) between 18 and 30 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kg (kilogram)
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of Merury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening and on Day -1
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including: Sinus rhythm, Pulse rate between 45 and 90 beats per minute (bpm), corrected QT (QTc) interval less than and equal to (<=) 450 millisecond (msec), QRS interval of <110 msec, PR interval less than (<) 200 msec. Morphology consistent with healthy cardiac conduction and function.
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, in addition to the user independent highly effective method of contraception, a man who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example [e.g.], condom with spermicidal foam/gel/film/cream/suppository) or must agree not to donate sperm, who is pregnant must use a condom.
* Non-tobacco user (nicotine substances, including tobacco products (e.g., cigarettes, e-cigarettes, cigars, chewing tobacco, gum or patch) (current and for past 6 months prior to screening)

Exclusion Criteria:

* Exposure to significant radiation for professional or medical reasons except dental x-rays (example, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to dosing. Exposure to X-rays of thorax and bone skeleton, (excluding spinal column) in the past 12 months
* Participants cannot have participated in a radiolabelled drug study for 12 months prior to dosing
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), syncope, hypotension, hypertension or vascular disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 milliLiter per minute (mL/min), kidney or urinary tract disturbances, thyroid disease, neurologic disease, significant psychiatric disorder, epilepsy, or fits of unexplained black-outs, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, that in the opinion of the investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence)
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen (325 milligram [mg]), within 14 days before the first dose of the study drug is scheduled until completion of the study
* Received a known inhibitor of cytochrome P450 (CYP) 3A4 or CYP2C9 activity within 28 days or a period less than 5 times the drug's half life (t1/2), whichever is longer, before the dose of the study drug is scheduled until completion of the study
* Received a known inducer of CYP3A4 or CYP2C9 activity within 28 days before the dose of study drug is scheduled until completion of the study
* Consumption of grapefruit products within 28 days before the first dose of the study drug is scheduled until completion of the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half life (t1/2), whichever is longer, before the dose of the study drug is scheduled
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 1 year before screening or positive test result(s) for alcohol, cotinine, and/or drugs of abuse (such as hallucinogens, barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and Day -1 of the treatment period
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 milliLitre [mL]) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* If a man, who plans to father a child while enrolled in the study or for 3 months after receiving the last dose of study drug
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies
* Regular use of tobacco or nicotine containing products in the past 6 months, as determined by medical history or participant's verbal report
* Positive test result(s) for nicotine at screening or Day -1 of the treatment period
* Recent changes in bowel habits (frequency, consistency, and amount) and irregular defecation pattern (less than one defecation per day)
* Preplanned surgery or procedures that would interfere with the conduct of the study
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator or employees of Johnson & Johnson
* Any participant who, in the opinion of the Investigator, should not participate in this study
* Has suicidal ideation with some intent to act, as per Columbia Suicide Severity Rating Scale (C-SSRS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time to Last Observed Quantifiable Concentration (T[last]) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The T(last) is the time to last observed quantifiable concentration.
Area Under the Curve From Time Zero to End of Dosing Interval (AUC[last]) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The AUC(last) is the measure of the plasma drug concentration from time zero to time of the last observed quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The AUC(infinity) is the area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Percent of AUC(0-infinity) Extrapolated (%AUC_extrap) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The %AUC_extrap is the percentage of AUC(0-infinity) accounted for by extrapolation. It is calculated as (AUC [infinity] minus [-] AUC[last])*100/ AUC[infinity], where AUC[infinity] is area under the plasma concentration versus time curve from time zero to extrapolated infinite time and AUC(last) is area under the plasma concentration time-curve from zero to the last measured concentration.
Elimination Half-Life (t[1/2]) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  The elimination half-life (t[1/2]) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Elimination Rate Constant (Lambda [z]) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Total Clearance (CL/F) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vd/F) | Predose (-0.5 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 32, 36, 48, 54, 60, and 72 hours postdose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vd/F) is influenced by the fraction absorbed.
Amount of Drug Excreted in Urine (Ae) | Up to Day 14
  Ae refers to the total amount of drug excreted in urine.
Percentage of Drug Excreted in Urine (%Ae) | Up to Day 14
  The %Ae is the percentage of drug dose excreted into the urine calculated as (Ae divided by dose)∗100.
Renal Clearance (CLr) | Up to Day 14
  The CLr is the renal clearance of the drug, calculated as Ae/AUC(0-infinity).
Amount of Drug Excreted in Feces (Fe) | Up to Day 14
  The Fe refers to the total amount of drug excreted in feces.
Percentage of Drug Excreted in Feces (%Fe) | Up to Day 14
  The %Fe is the total amount excreted in feces, expressed as a percentage of the administered dose.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | From Screening to End of study (Approximately up to 46 days)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Madison, Wisconsin, United States